CLINICAL TRIAL: NCT05940922
Title: Characteristics, ImmunoglobulinTreatment Patterns, and Effectiveness in CIDP, Heredofamilial Amyloidosis, and Guillain-Barré Syndrome
Brief Title: RWE-based Treatment Patterns and Outcomes in CIDP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RwHealth (Industry)
Collaborators: Alnylam Pharmaceuticals (Industry); Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RWH_LS_CIDPv2
Record Dates: First submitted 2023-05-22; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; Guillain-Barre Syndrome; Hereditary Amyloidosis
Keywords: Inflammatory polyneuropathies
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Guillain-Barre Syndrome; Amyloidosis, Familial; Neuritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIDP GBS hATTR: Adult patients diagnosed and treated at the study centre for chronic inflammatory demyelinating polyneuropathy (CIDP), or Guillain-Barre syndrome (GBS), or heredofamilial amyloidosis (hATTR).
  Interventions: Other: No intervention. Retrospective observation only.

INTERVENTIONS:
Other: No intervention. Retrospective observation only. — No intervention. Retrospective observation only.

SUMMARY:
To describe the demographics, clinical characteristics, treatment patterns and clinical outcomes of chronic inflammatory demyelinating polyneuropathy (CIDP), Guillain-Barre Syndrome (GBS), and heredofamilial amyloidosis (hATTR) adult patients at a single U.K. centre.

DETAILED DESCRIPTION:
CIDP (chronic inflammatory demyelinating polyneuropathy) is an immune-mediated peripheral nerve disorder, that can be progressive or relapsing, with sensory or motor symptoms. It is typically diagnosed by a combination of progressive history, ruling out other neuropathic conditions, or by being refractive to immunoglobulin or corticosteroid treatment. Recently published guidelines introduced a pathway to diagnosis (Van den Burgh, 2021). Challenges with CIDP can result in misdiagnoses of hereditary amyloidosis (hATTR) and Guillain-Barré syndrome (GBS).

Studies in France, Italy, and Japan indicate that 15-53% of patients with hereditary amyloidosis (hATTR) have previously been diagnosed with CIDP (Russo 2020; Cortese 2017; Plante-Bordeneuve 2007; Koike 2011).

A study in the Netherlands highlighted the diagnostic challenges in diagnosis of acute onset CIDP versus (GBS) during the early acute phase onset (Ruts 2010). This diagnostic challenge may be driven by the lack of diagnostic tests or clinical features that can distinguish GBS acute onset CIDP (Van den Burgh, 2021).

A Hospital, Episode Statistics (HES) analysis of previous and subsequent primary diagnosis codes for CIDP patients highlighted hATTR and GBS, as well as unspecified [inflammatory] neuropathy codes, as three conditions with diagnostic challenges that might lead to reclassification of patients.

This current study is designed to describe the real-world demographics, clinical characteristics, and treatment pathways of patients diagnosed with CIDP, GBS and hATTR. In addition, this study will describe the real-world effectiveness and safety of immunoglobulin therapies in the treatment of patients with CIDP or GBS.

2.2. Objectives Primary Objective: To describe the baseline demographic and clinical characteristics CIDP, GBS and hATTR patients at a single U.K. centre, part of the Northern Care Alliance NHS Trust, in order to improve the understanding of the natural history of these neuropathic diseases.

Secondary Objectives:

* Describe the Ig treatment pathway and treatment-related outcomes in CIDP patients.
* Compare the Ig treatment pathway and treatment-related outcomes between typical and atypical CIDP
* Describe the characteristics of CIDP patients who are refractory to Ig treatment.

2.3. Study design This is a non-interventional, retrospective observational cohort study using the data collected during routine clinical appointments of patients with CIDP, hATTR, or GBS attending the Northern Care Alliance NHS Trust.

There will be no additional data collection or additional interventions carried out as part of this study.

All NHS patients have the opportunity to "opt out" as part of the national data opt-out is a service that allows patients to opt out of their confidential patient information being used for research and planning. Only data from patients who did not "opt out" will be used.

2.4. Population CIDP, GBS, and hATTR patients aged 18 years or over at diagnosis. 2.5. Variables

* CIDP, GBS and hATTR patient identifiers
* Demographics and clinical characteristics
* Treatments prescribed, with a focus on immunoglobulins and corticosteroids
* Clinical outcomes (grip strength test; 9-hole peg test; 50m walk test; Berg balance).

See section 4, table 2 for complete variable list. 2.6. Data sources Electronic medical records including inpatient, outpatient pharmacy datasets. The Ig Database dataset: NHS database of immunoglobulin therapy use, in which treatment data (date/dose) as well as outcome measures for patients who have received immunoglobulin therapy are recorded. This database is supported by MD-SAS.

3. Research question, objectives, and endpoints 3.1. Primary objectives To describe the demographics and clinical characteristics of CIDP, hATTR, and GBS patients in a single centre in the North West of England.

3.2. Primary endpoints

• Summary statistics and distributions of patient demographics reported for all patients diagnosed with CIDP, hATTR, or GBS, and by relevant subgroups, including:

* Age at diagnosis of CIDP, hATTR, or GBS
* Sex
* Ethnicity
* Comorbid diabetes
* CIDP type: typical, variant (distal, multifocal, focal, motor, sensory).
* Presenting symptoms at diagnosis
* History of [bilateral] carpel tunnel syndrome
* Genetic testing (for hATTR)
* Antibody testing IgM/IgG:
* Anti-neurofascin 155 (anti-NF155)
* Anti-contactin 1 (anti-CNTN1
* CIDP effectiveness measures at diagnosis or pre-Ig treatment initiation:
* Grip strength test (mean and range)
* 9-hole peg test (mean and range)
* 10m walk test (mean and range)
* Berg balance test (mean and range)
* Overall neuropathy limitations scale
* Medical research council muscle strength score
* Referrals to external centres

3.3. Secondary objectives

There are several secondary objectives:

* To describe the diagnostic pathways of CIDP, hATTR, and GBS patients in a single centre in the North West of England.
* To describe the effectiveness of intravenous and/or subcutaneous immunoglobulin in CIDP and GBS patients in a real-world setting in a single centre in the in the North West of England and nationally using the NHS Ig Database.
* To describe the treatment patterns of intravenous and/or subcutaneous immunoglobulin in CIDP and GBS patients in a real-world setting in a single centre in the in the North West of England and nationally using the NHS Ig Database.

3.4. Secondary endpoints

* For each confirmed CIDP, GBS and hATTR patient at the single centre in the North West: list the previous neurological diagnosis codes (see Table 1) recorded in EHR, and frequency of previous codes (e.g. 1, 2, 3 or more.)
* For confirmed CIDP and GBS patients receiving immunoglobulin and present in the NHS Ig Database: record the changes in the following measurement outcomes taken prior to treatment start and at the end (~8 weeks later), stratified by patient demographics, clinical characteristics, and treatment:
* For confirmed CIDP and GBS patients receiving Ig and present in the NHS MD-SAS database, stratified by patient demographics, clinical characteristics, and treatment:
* Time from diagnosis to start of Ig treatment
* Proportion of patients receiving IV or SC at start of treatment
* Proportion of patients switching from IV to SC, or SC to IV
* Proportion of patients receiving Ig under homecare, stratified by IV or SC
* Median duration and range of each cycle of Ig treatment.
* Median time to Ig dose tapering.
* Percentage of Ig-treated patients who do not respond to treatment
* Percentage of Ig-treated patients who discontinue therapy, stratified by reason for discontinuation.
* Frequency of patients that achieve remission after each cycle of Ig treatment:
* Never
* A least once.
* 2-5 times.
* 5+ times.
* Median duration and range of remission.
* Relapse-free survival (where T0 is the last recorded Ig treatment): median and range.
* Frequency of relapse [set time duration: ever, in the last 12 months, 2 years, 5 years, 5+ years]:
* Never
* A least once.
* 2-5 times.
* 5+ times.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed or treated at the study centre with a diagnosis of chronic inflammatory demyelinating polyneuropathy (CIDP), Guillain-Barre syndrome (GBS), or heredofamilial amyloidosis (hATTR).
* Patients aged 18 years and over.
* Patients who did not "opt out" of their health data being used for research.

Exclusion Criteria:

• Patients who "opted out" of their health data being used for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective medical data review of patients diagnosed with chronic inflammatory demyelinating polyneuropathy (CIDP), Guillain-Barre syndrome (GBS), or heredofamilial amyloidosis (hATTR) at a single centre in the United Kingdom, and who received immunoglobulin treatment.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-08-17 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Patient baseline characteristics | At diagnosis
  Patient demographics, clinical characteristics, weight (kg), and medical history.
Grip strength test | At diagnosis or pre-Ig treatment initiation.
  Average measurement of grip strength using dynamometer over 3 trials per hand, measured in kilograms of force.
9-hole peg test | At diagnosis or pre-Ig treatment initiation.
  Average of four measurements (two per hand) in seconds, measured using stopwatch.
10 meter walk test | At diagnosis or pre-Ig treatment initiation.
  Average speed in meters/second over 10 meters, measured using stopwatch.
Overall neuropathy limitations scale | At diagnosis or pre-Ig treatment initiation.
  The ONLS allows semi-objective measurement of function, which is useful to detect changes with therapy, and relatively earlier changes may be detected than on the standard five-point Medical Research Council scale used in routine examination of muscle power.
  The ONLS is graded separately for upper and lower limbs as follows:
  Arm scale score (0 to 5) + Leg scale score (0 to 7) for the total out of 12.
Berg balance test | At diagnosis or pre-Ig treatment initiation.
  The Berg balance uses a stopwatch, a ruler or a measuring tape, a chair, a step, and an object that can be picked up. It takes ~15 min to complete and includes 14 tasks scored 0-4 and scores are added for a total out of 56.
  Berg balance test scoring system:
  0 to 20: Score - need the assistance of a wheelchair to move around safely 21 to 40: Score - need some type of walking assistance, cane or a walker 41 to 56: Score - considered independent and able to move around safely without assistance
Medical research council muscle strength score | At diagnosis or pre-Ig treatment initiation.
  The Medical Research Council (MRC) Scale for Muscle Strength is a commonly used scale for assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction)
  The Criteria requires that each of the six muscle groups listed below are examined bilaterally, each with a score from 0 to 5 according to the scale:
  Shoulder abductors, Elbow flexors, Wrist extensors, Hip flexors, Knee extensors, Foot dorsiflexors.
Inflammatory neuropathy cause and treatment (INCAT) sensory sum (ISS) score | At diagnosis or pre-Ig treatment initiation up to December 31, 2022 or death or lost-to-follow-up, whichever comes first.
  The ISS score is inversely related to function, with 0 representing no functional impairment and 10 representing inability to make any purposeful movement with either arms or legs.

SECONDARY OUTCOMES:
Time to treatment initiation | From diagnosis to day 1 of treatment
  Time to start of immunoglobulin treatment in CIDP patients, measured in days.
Treatment patterns | From the date of first immunoglobulin up to December 31, 2022 or death or lost-to-follow-up, whichever comes first.
  Describe the frequency (number of immunoglobulin treatments per year), the median duration (months), and dosing of immunoglobulin therapy (cumulative g/kg) in CIDP patients.
Treatment outcomes | Treatment outcomes to be measured at 6 week intervals after the date of first immunoglobulin up to December 31, 2022 or death or lost-to-follow-up, whichever comes first.
  Establish the frequency of patients who achieved remission, stable disease, or did not respond to immunoglobulin treatment.
Relapse | From 6 weeks after the date of first immunoglobulin treatment to the date of first documented relapse up to a maximum of 173 months of follow-up
  Describe frequency of relapse and median relapse-free survival in CIDP patients treated with immunoglobulin. A CIDP relapse is defined as a deterioration (ie, increase) by at least 1 point in the total ISS score (range 0 [healthy] to 10 [unable to make any purposeful movements with arms or legs]) at any treatment visit after treatment initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Care Alliance NHS Foundation Trust, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: No